CLINICAL TRIAL: NCT06919432
Title: Efficacy of Triple-daily 15mA Transcranial Alternating Current Stimulation on Adolescent Non-suicidal Self-injury (NSSI): a Double-blind, Randomized, Sham-controlled Trial
Brief Title: Efficacy of Triple-daily 15mA tACS on Adolescent NSSI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Principal Investigator, Tianhong ZHANG, Associate Professor, Shanghai Mental Health Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024y1023
Record Dates: First submitted 2025-04-02; First posted 2025-04-09 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Self-Injurious Behavior
Keywords: Transcranial Alternating Current Stimulation (tACS); non-invasive brain stimulation
MeSH Terms: conditions — Self-Injurious Behavior

STUDY DESIGN:
Intervention Model Description: The present clinical protocol is designed as a double-blind, parallel, sham-controlled, randomized clinical trial.
Who Masked: Participant, Outcomes Assessor
Masking Description: Both clinical staff and participants were blinded to the assignment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the active-tACS group (Experimental): This trial consists of a 2-week intensified intervention phase (40 sessions), followed by a 4-week observation period. On the first day of the intervention, participants will receive a tACS session, followed by triple-daily tACS sessions administered for 13 consecutive days.
  Interventions: Device: Active-tACS
- the sham-tACS group (Sham Comparator): Participants in the sham-tACS group will undergo the same protocol, utilizing a sham tACS incapable of delivering active stimulation. They will be kept unaware of their assigned treatment.
  Interventions: Device: Sham-tACS

INTERVENTIONS:
Device: Active-tACS — Participants were comfortably positioned on a lounge chair and received alternating current stimulation using an FDA-approved tACS device (Nexalin Technology, Inc., Houston, TX, USA). Electrodes were evenly placed across the forehead and mastoid regions. Trained nurses administered the tACS according to standardized protocols.
  Arms: the active-tACS group
Device: Sham-tACS — The sham tACS device will resemble the active stimulation device in appearance, weight, size, color, and odor, ensuring indistinguishability for the patients. Throughout the entire intervention period, each participant will be allocated to the same tACS device, regardless of whether it delivers active or sham stimulation.
  Arms: the sham-tACS group

SUMMARY:
In order to assess the clinical efficacy of triple-daily 15mA-tACS stimulation by comparing the effects of active and sham tACS interventions on driving improvements in adolescent Nonsuicidal Self-Injury(NSSI), participants will be randomly assigned to either the active or sham tACS group. This trial consists of a 2-week intensified intervention phase (40 sessions), followed by a 4-week observation period. The key hypothesis is that triple-daily 15mA-tACS stimulation will enhance clinical recovery compared to sham stimulation.

DETAILED DESCRIPTION:
Recognizing the clinical shortcomings of traditional methods for adolescent NSSI, study objective is to establish evidence supporting the efficacy of a triple-daily 15mA-tACS stimulation regimen targeting the forehead and both mastoids. This intervention will be administered five days a week over a four-week treatment period, with the aim of eliciting substantial clinical improvements in adolescent NSSI compared to a sham intervention. On the first day of the intervention, participants will receive a tACS session, followed by triple-daily tACS sessions administered for 13 consecutive days. Following the completion of treatment, participants will undergo follow-up observations every 7 days for 4 weeks. EEG and ECG recordings will be obtained at baseline, on day 1 after the first session, at the end of the 2-week intervention period (after 40 sessions), and at the 6-week follow-up. Throughout the sessions, all evaluations will be conducted under standardized conditions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of NSSI based on the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria section 3 diagnostic criteria.
* Five or more NSSI episodes in the past year and at least one NSSI episode in the past month.
* Age between 12 and 21 years.
* Informed consent from parents or legal guardians.
* Informed consent from participants aged 15 years and above.

Exclusion Criteria:

* Current or history of organic brain disorders or neurological disorders.
* Elevated or imminent suicidal risk, as assessed by clinicians during routine screening.
* Previous or current exposure to electroconvulsive therapy (ECT), modified ECT, TMS, transcranial direct current stimulation (tDCS), tACS, or other neurostimulation treatments.
* Presence of cochlear implants, cardiac pacemakers, implanted devices, or metal in the brain.
* Previous or current use of psychotropic medication.
* Pregnancy or lactation.
* Participation in another concurrent clinical trial.
* Refusal to provide informed consent to participate in the trial.
* Other circumstances deemed unsuitable for participation by researchers.

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in total NSSI incidents during the 4-week follow-up period post-intervention | 6 weeks
  It will be determined by the Suicide and Self-Injury Behavior Interview-Revised (SITBI-R). The primary outcome is the proportion of participants achieving a ≥50% decrease in NSSI frequency within the past month at Day 42, as measured by the SITBI-R. A threshold of 50% reduction was selected based on its clinical relevance as an indicator of intervention efficacy.
Change in mean NSSI severity levels during the 4-week follow-up period post-intervention | 6 weeks
  It will be determined by the Suicide and Self-Injury Behavior Interview-Revised (SITBI-R). The SITBI-R assesses NSSI severity using a 5-point scale (minimum = 1, maximum = 5), where higher scores indicate more severe outcomes: Level 1 (mild NSSI without skin damage) to Level 5 (severe NSSI requiring medical intervention). Comparative analysis of severity-level changes between the active-tACS and sham-tACS groups will be conducted at the 4-week follow-up post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: TianHong Zhang, Doctor, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No